CLINICAL TRIAL: NCT03193593
Title: Phase 2 Placebo-Controlled, Double Blind, Ascending Dose Cohort Study to Evaluate Safety and Efficacy of EB-001 IM Injections in Reducing Musculoskeletal Pain in Subjects Undergoing Elective Augmentation Mammoplasty (Breast Augmentation)
Brief Title: Study to Evaluate EB-001 in Reducing Musculoskeletal Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bonti, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EB001-MA201
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Placebo Injections (Placebo Comparator): Intervention: Drug: Placebo
  Single Saline Injection into the Pectoralis Muscle
  Interventions: Drug: Placebo
- EB-001 Dose 1 (Active Comparator): Intervention: Drug: EB-001
  1st Dose in escalation paradigm. Single Injection of active drug into the pectoralis muscle
  Interventions: Drug: EB-001
- EB-001 Dose 2 (1.6X) (Active Comparator): Intervention: Drug: EB-001
  2nd Dose in escalation paradigm, 1.6X Dose 1. Single Injection of active drug into the pectoralis muscle
  Interventions: Drug: EB-001
- EB-001 Dose 3 (3.3X) (Active Comparator): Intervention: Drug: EB-001
  3rd Dose in escalation paradigm, 3.3X Dose 1. Single Injection of active drug into the pectoralis muscle
  Interventions: Drug: EB-001
- EB-001 Dose 4 (6.7X) (Active Comparator): Intervention: Drug: EB-001
  4th Dose in escalation paradigm, 6.7X Dose 1. Single Injection of active drug into the pectoralis muscle
  Interventions: Drug: EB-001
- EB-001 Dose 5 (10X) (Active Comparator): Intervention: Drug: EB-001
  5th Dose in escalation paradigm, 10X Dose 1. Single Injection of active drug into the pectoralis muscle
  Interventions: Drug: EB-001
- EB-001 Dose 6 (13.3X) (Active Comparator): Intervention: Drug: EB-001
  6th Dose in escalation paradigm, 13.3X Dose 1. Single Injection of active drug into the pectoralis muscle
  Interventions: Drug: EB-001

INTERVENTIONS:
Drug: Placebo — Placebo- Single injection of saline into Pectoralis Muscle
  Arms: Placebo Injections
Drug: EB-001 — Single injection of EB-001 into Pectoralis Muscle
  Arms: EB-001 Dose 1; EB-001 Dose 2 (1.6X); EB-001 Dose 3 (3.3X); EB-001 Dose 4 (6.7X); EB-001 Dose 5 (10X); EB-001 Dose 6 (13.3X)

SUMMARY:
To determine the safety and efficacy of single intra-operative treatment of EB-001 IM injections into the Pectoralis Major (PM) in subjects undergoing breast augmentation with subpectoral implants

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of EB-001 in decreasing post-surgical pain in patients undergoing surgical breast augmentation with subpectoral placement of the implants. Intramuscular (IM) injection of EB-001 into the PM bilaterally during surgery may decrease pain related to stretching of the PM by the implants.

The safety objective is to determine the safety and tolerability of single intraoperative treatment of EB-001 IM injections into the PM in subjects undergoing breast augmentation with subpectoral implants.

The efficacy objective is to evaluate the efficacy of intraoperative administration of EB-001 IM into the PM in reducing the pain and use of rescue pain medications in subjects undergoing breast augmentation with subpectoral implants.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 to 55 years of age, inclusive
2. Women who are in good health as determined by medical history, physical examination, clinical laboratory studies, ECGs, vital signs, and Investigator judgment
3. Scheduled to undergo primary breast augmentation under general anesthesia (endotracheal or otherwise) with:

   1. Sub-pectoral implants placement,
   2. Infra-mammary surgical approach,
   3. Implant size between 250 and 400cc and
   4. Non-textured saline breast implants
4. American Society of Anesthesiologist (ASA) Physical Class 1-2
5. Women of non-childbearing potential or postmenopausal (at least 12 consecutive months of amenorrhea)
6. Women of childbearing potential must not be pregnant, lactating, or planning to become pregnant during the study
7. Women of childbearing potential agreeing to use either:

   1. a highly effective method of contraception with failures rates less than 1% per year such as implant, intrauterine device (IUD), or confirmed sterilization and sterilization procedure at least 3 months prior to the day of dosing
   2. dual methods of contraception with overall failures rate less than 1% per year such as injectable, pill, patch, ring, and diaphragm from the day of dosing for 3 months (subjects using oral contraception must have initiated treatment at least 2 months prior to the day of dosing)
8. Willing and able to complete protocol requirements and instructions, which includes completion of all required visits, procedures and in-clinic stays until the end of the study
9. Willing and able to sign and date IRB-approved informed consent
10. Able to speak, read, and understand the language of the informed consent form (ICF) and study questionnaires

Exclusion Criteria:

1. History of surgical procedure involving the breast, including, but not limited to, breast augmentation. History of minor localized breast biopsy is not exclusionary if it occurred at least 1 year prior to the screening visit, and if considered not clinically significant in the opinion of the investigator.
2. Pre-existing lung disease that could impact subject safety in the opinion of the investigator
3. History of smoking within the past two years
4. Slow vital capacity that is below 80% of normal value for respective race, age, height, and gender
5. Pulse oximetry below 95%
6. Body weight less than 50 kg (110 pounds) or a Body Mass Index (BMI) of ≥ 32
7. Documented diagnosis of chronic pain condition, or other painful pre-operative condition that, in the opinion of the investigator, may require analgesic treatment in the post-operative period (e.g. significant joint pain, neuropathic pain)
8. Known hypersensitivity to any botulinum toxin serotype or to any component of the formulation
9. Reported use of any botulinum toxin within 3 months prior to the date of surgery
10. Anticipated use of any botulinum toxin of any serotype during the study
11. Use of long acting opioids within 3 days or any opioid medication within 24 hours prior to surgery
12. Aminoglycoside intake within 48 hours prior to or during surgery
13. Pre-existing disorders of the neuromuscular junction (myasthenia gravis, Eaton- Lambert syndrome, or amyotrophic lateral Sclerosis)
14. Any past or current medical condition that in opinion of investigator, puts subject at undue safety risk for surgical complications or for use of the investigational product.
15. Any clinically significant psychiatric condition that, in opinion of investigator, may interfere with study assessments or protocol compliance
16. History of alcohol or drug abuse in the last 3 years, based on investigator judgement
17. Current enrollment in an investigational drug or device study or participation in such a study within 30 days or 5 half-lives of the drug, whichever is longer, of entry into this study
18. Subject plans to donate blood or plasma from 30 days prior to screening until last follow-up visit (Day 29)
19. Reported pain score of 2 or more at screening on the 11-point scale NPRS-A following strength testing with PM activation

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-08-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lotus Clinical Research, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Injections: Placebo Injection into the Pectoralis Muscle
- EB-001 Dose 1 (1X): 1st Dose in escalation paradigm.
  Injection of active drug into the pectoralis muscle
- EB-001 Dose 2 (1.6X): 2nd Dose in escalation paradigm, 1.6X Dose 1.
  Injection of active drug into the pectoralis muscle.
- EB-001 Dose 3 (3.3X): 3rd Dose in escalation paradigm, 3.3X Dose 1.
  Injection of active drug into the pectoralis muscle.
- EB-001 Dose 4 (6.7X): 4th Dose in escalation paradigm, 6.7X Dose 1.
  Injection of active drug into the pectoralis muscle.
- EB-001 Dose 5 (10X): 5th Dose in escalation paradigm, 10X Dose 1.
  Injection of active drug into the pectoralis muscle.
- EB-001 Dose 6 (13.3X): 6th Dose in escalation paradigm, 13.3X Dose 1.
  Injection of active drug into the pectoralis muscle.
Period: Overall Study
Arm/Group | Placebo Injections | EB-001 Dose 1 (1X) | EB-001 Dose 2 (1.6X) | EB-001 Dose 3 (3.3X) | EB-001 Dose 4 (6.7X) | EB-001 Dose 5 (10X) | EB-001 Dose 6 (13.3X)
Started | 18 | 4 | 4 | 4 | 8 | 16 | 12
Completed | 14 | 3 | 3 | 4 | 7 | 13 | 8
Not Completed | 4 | 1 | 1 | 0 | 1 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- EB-001 Dose 1 (1X): 1st Dose in escalation paradigm.
  Single Injection of active drug into the pectoralis muscle
- EB-001 Dose 2 (1.6X): 2nd Dose in escalation paradigm, 1.6X Dose 1.
  Single Injection of active drug into the pectoralis muscle.
- EB-001 Dose 3 (3.3X): 3rd Dose in escalation paradigm, 3.3X Dose 1.
  Single Injection of active drug into the pectoralis muscle.
- EB-001 Dose 4 (6.7X): 4th Dose in escalation paradigm, 6.7X Dose 1.
  Single Injection of active drug into the pectoralis muscle.
- EB-001 Dose 5 (10X): 5th Dose in escalation paradigm, 10X Dose 1.
  Single Injection of active drug into the pectoralis muscle.
- EB-001 Dose 6 (13.3X): 6th Dose in escalation paradigm, 13.3X Dose 1.
  Single Injection of active drug into the pectoralis muscle.
- Total: Total of all reporting groups
Arm/Group | Placebo Injections | EB-001 Dose 1 (1X) | EB-001 Dose 2 (1.6X) | EB-001 Dose 3 (3.3X) | EB-001 Dose 4 (6.7X) | EB-001 Dose 5 (10X) | EB-001 Dose 6 (13.3X) | Total
Number analyzed (Participants) | 18 | 4 | 4 | 4 | 8 | 16 | 12 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (4.66) | 29.5 (4.36) | 28.8 (6.08) | 27.0 (3.37) | 27.3 (4.30) | 27.3 (3.14) | 27.3 (3.14) | 27.6 (3.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 4 | 4 | 4 | 8 | 16 | 12 | 66
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 2 | 1 | 1 | 3 | 1 | 6 | 21
  White | 10 | 2 | 3 | 3 | 5 | 14 | 5 | 42
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 4 | 4 | 4 | 8 | 16 | 12 | 66
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 22.57 (2.596) | 23.95 (2.958) | 23.00 (3.614) | 22.40 (2.848) | 22.66 (2.630) | 22.94 (2.117) | 23.18 (2.474) | 23.00 (2.437)

OUTCOME MEASURES:

1. Primary Outcome: Subject's Assessment of Pain Using the Numeric Pain Rating Scale (AUC16h-96h)
Description: Subject's assessment of pain using the Numeric Pain Rating Scale (1= No Pain, 10= Maximum Pain) for the first 96 hours following injection, expressed as AUC over the 16h to 96h period following dosing.
Time Frame: 16 hours to 96 hours following dosing
Population: mITT
Measure: Mean (Standard Deviation); unit: units on a Scale*hours
Arm/Group | Placebo Injections | EB-001 Dose 1 (1X) | EB-001 Dose 2 (1.6X) | EB-001 Dose 3 (3.3X) | EB-001 Dose 4 (6.7X) | EB-001 Dose 5 (10X) | EB-001 Dose 6 (13.3X)
Number analyzed (Participants) | 18 | 4 | 4 | 4 | 8 | 16 | 12
units on a Scale*hours | 289.18 (211.552) | 341.78 (124.655) | 401.75 (310.509) | 290.55 (224.966) | 333.44 (217.742) | 381.82 (199.401) | 340.89 (155.328)

ADVERSE EVENTS:
Time Frame: 30 Days
Arm/Group | Placebo Injections | EB-001 Dose 1 (1X) | EB-001 Dose 2 (1.6X) | EB-001 Dose 3 (3.3X) | EB-001 Dose 4 (6.7X) | EB-001 Dose 5 (10X) | EB-001 Dose 6 (13.3X)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/4 | 0/4 | 0/4 | 0/8 | 0/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/4 | 0/4 | 0/4 | 1/8 | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 15/18 | 3/4 | 4/4 | 4/4 | 7/8 | 14/16 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Injections (N=18) | EB-001 Dose 1 (1X) (N=4) | EB-001 Dose 2 (1.6X) (N=4) | EB-001 Dose 3 (3.3X) (N=4) | EB-001 Dose 4 (6.7X) (N=8) | EB-001 Dose 5 (10X) (N=16) | EB-001 Dose 6 (13.3X) (N=12)
Breast Hematoma (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Injections (N=18) | EB-001 Dose 1 (1X) (N=4) | EB-001 Dose 2 (1.6X) (N=4) | EB-001 Dose 3 (3.3X) (N=4) | EB-001 Dose 4 (6.7X) (N=8) | EB-001 Dose 5 (10X) (N=16) | EB-001 Dose 6 (13.3X) (N=12)
Nausea (Gastrointestinal disorders) | 13 (13) | 3 (3) | 3 (3) | 4 (4) | 6 (6) | 14 (14) | 6 (6)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 6 (6) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT03193593/Prot_SAP_000.pdf